CLINICAL TRIAL: NCT06621641
Title: Outcomes of a Nurse-led High-flow Nasal Cannula Weaning Protocol in Pediatric Critical Bronchiolitis Patients
Brief Title: Nurse-led High-flow Nasal Cannula Weaning Protocol in Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Hasan ağın, Prof. Doctor, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02024/GOA-80
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Bronchiolitis; Respiratory Failure (Pediatric Patients); High Flow Nasal Cannula
Keywords: bronchiolitis; high flow nasal cannula; Quality Improvement (QI); HFNC protocol
MeSH Terms: conditions — Bronchiolitis; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled trial will be conducted to evaluate the effectiveness of a newly developed HFNC (High-Flow Nasal Cannula) weaning protocol in infants aged 1-24 months with bronchiolitis, compared to the standard weaning protocol.
  Participants:
  Infants aged 1-24 months admitted with bronchiolitis and receiving HFNC therapy will be included. Exclusion criteria include infants born before 32 weeks of gestation or those with cardiopulmonary, genetic, congenital, or neuromuscular abnormalities.
  Randomization and Groups:
  Participants will be randomly assigned to one of two groups:
  Control Group: Will follow the existing HFNC weaning protocol. Intervention Group: The intervention group will follow the newly developed multidisciplinary HFNC weaning protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Protocol Group (No Intervention): Control Arm (Pre-Protocol Implementation):
  This group includes patients aged 1-24 months receiving HFNC (High-Flow Nasal Cannula) therapy for bronchiolitis based on the conventional, non-standardized approach. HFNC weaning decisions in this group are made at the treating clinicians' discretion, without following a formal protocol. Decisions are influenced by clinical presentation, respiratory effort, and clinician experience. This group serves as the control arm, representing the current standard of care.
- New Protocol Group (Active Comparator): This group includes patients aged 1-24 months who are randomized to receive HFNC therapy under a newly implemented standardized weaning protocol, developed using Quality Improvement (QI) methodology. The protocol involves a structured, criteria-based weaning approach with clear steps for reducing HFNC support, focusing on clinical indicators like respiratory rate, work of breathing, and oxygen saturation. A multidisciplinary team, including pediatricians, nurses, and respiratory therapists, created this protocol, and staff received training before implementation.
  Interventions: Behavioral: The new HFNC weaning protocol

INTERVENTIONS:
Behavioral: The new HFNC weaning protocol — Patients will be randomly assigned to two groups: one following the new HFNC weaning protocol and another using the standard care protocol. The new protocol includes stepwise flow reduction based on the patient's clinical stability and uses the Respiratory Assessment Scale (RAS) to monitor weaning progress. The protocol emphasizes a multidisciplinary approach involving pediatricians, nurses, and respiratory therapists, with consistent training and application of weaning criteria
  Arms: New Protocol Group

SUMMARY:
Bronchiolitis is a leading cause of pediatric hospital admissions. Despite its limited clinical benefits, the use of HFNC in children with bronchiolitis is increasing.

Previous studies using quality improvement (QI) methodologies have successfully reduced HFNC usage through weaning protocols and trials of standard oxygen therapy.

This study involves implementing an HFNC initiation and weaning protocol at Aydın Maternity and Children's Hospital, involving infants aged 1-24 months admitted with bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis is a leading cause of pediatric hospital admissions. While high-flow nasal cannula (HFNC) is effective as a rescue therapy for patients with severe respiratory distress when standard oxygen therapy fails, studies suggest that early use of HFNC in moderate cases does not significantly improve outcomes such as hospital stay duration or intubation rates. Despite its limited clinical benefits, the use of HFNC in children with bronchiolitis is increasing, raising concerns about unnecessary treatment and extended hospital stays due to a lack of standardized weaning protocols.

Evidence suggests that HFNC should be used effectively as a rescue treatment after standard oxygen therapy fails, serving as an intermediate step before invasive support. However, the high costs and self-limiting nature of bronchiolitis necessitate reducing the overuse of HFNC in hospitalized children. Previous studies using quality improvement (QI) methodologies have successfully reduced HFNC usage through weaning protocols and trials of standard oxygen therapy.

This study involves implementing an HFNC initiation and weaning protocol at Aydın Maternity and Children's Hospital, involving infants aged 1-24 months admitted with bronchiolitis. A multidisciplinary team will evaluate patients using the Respiratory Assessment Scale (RAS), with mild, moderate, and severe classifications. The study compares HFNC duration, hospital stay, oxygen support duration, and associated costs before and after the protocol implementation.

Exclusion Criteria:

Premature infants born at less than 32 weeks Patients with cardiopulmonary, genetic, congenital, or neuromuscular abnormalities were excluded.

A prospective, randomized controlled trial will be conducted to evaluate the effectiveness of a newly developed HFNC (High-Flow Nasal Cannula) weaning protocol in infants aged 1-24 months with bronchiolitis, compared to the standard weaning protocol.

The new HFNC weaning protocol was developed using Quality Improvement (QI) methodology, involving input from pediatricians, nurses, and hospital staff through training sessions. The training lasted one month before the implementation, focusing on classifying patients using the Respiratory Assessment Scale (RAS), which includes respiratory rate, the workload of breathing, and consciousness level. A multidisciplinary team will apply the protocol.

Protocol for Bronchiolitis in Children Under 2 Years:

Aspiration, postural drainage, hydration, antipyretics if necessary, nasal cannula for SpO₂ drop (3-4 L/min)

Despite nasal cannula >3 LPM (FiO₂: 32), hypoxemia (≤92% FiO₂) or moderate-to-severe RAS:

Yes: Start HFNC (High-Flow Nasal Cannula) therapy. No: Continue with HFNC or nasal cannula/mask.

HFNC Therapy Initiation:

Initial FiO₂: 50%, Flow rate: 1-2 L/kg Target SpO₂ between 92-96% by titrating FiO₂. Calculate the baseline ROX index.

Reassess in 30-60 minutes:

Is there clinical deterioration? (Moderate-to-severe RAS)

If clinical deterioration is present:

FiO₂ ≥ 50% SpO₂ < 90% pCO₂ ≥ 60 Positive pressure ventilation should be considered if there is apnea or bradycardia.

If there is no clinical deterioration:

After 4 hours of stable condition, reassess. Is there improvement in RAS and ROX index, and is the patient clinically stable?

Yes:

If FiO₂ < 30%, start weaning the flow rate and FiO₂ simultaneously. Reduce the flow rate by 2 L/min every 2-4 hours, and evaluate the RAS-ROX trend every 2-4 hours.

If there is respiratory deterioration:

Continue or increase HFNC flow rate and FiO₂ as needed.

If there is no respiratory deterioration:

Weaning continues. Discontinue HFNC when the flow rate reaches 4 L/min and FiO₂ < 30%.

Is there respiratory deterioration?

Yes:

Return to the previous flow rate, and reassess within 30 minutes.

Randomization and Groups:

Participants will be randomly assigned to one of two groups:

Control Group: Will follow the existing HFNC weaning protocol. Intervention Group: The intervention group will follow the newly developed multidisciplinary HFNC weaning protocol.

Outcomes:

The 2 groups will be compared regarding HFNC duration, hospital stay, oxygen support duration, intensive care readmission, noninvasive ventilation (NIV) needs, intubation rates, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 1 month and younger than 24 months of age; hospitalized at the PICU with the intention of treatment with HFNC at least for the upcoming 4 hours
* Patients with moderate and severe RAS(Respiratory Assessment Scale) requiring HFNC
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation

Exclusion Criteria:

* İnfants born before 32 weeks of gestation or those with cardiopulmonary, genetic, congenital, or neuromuscular abnormalities.
* Patient with an indication for immediate noninvasive ventilation (NIV)
* Patients deemed at high risk for the need for non-invasive mechanical ventilation within the next 4 hours
* Hemodynamic instability

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
HFNC duration | Through study completion, an average of 1 year
  HFNC duration calculated during intensive care hospitalization
Hospital length of stay | Through study completion, an average of 1 year
  Total hospital stay time including intensive care unit
Need for non-invasive ventilation | Through study completion, an average of 1 year
  It will be compared whether there is a difference between the two groups in terms of niv needs.
Associated costs | Through study completion, an average of 1 year
  HFNC costs and total hospitalization costs will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Prof.Dr., Study Chair — Dr. Behcet Uz Children's Hospital
Locations (6):
- Turkey (Türkiye) (6):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Erzurum Regional Research and Training Hospital, Erzurum
  - Cam Sakura Research and Training Hospital, Istanbul
  - Acibadem University, Acibadem Altunizade Hospital, Istanbul
  - Istanbul Aydin University, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang JX, Colwell B, Vadlaputi P, Sauers-Ford H, Smith BJ, McKnight H, Witkowski J, Padovani A, Aghamohammadi S, Tzimenatos L, Beck Rn S, Reneau K, Nill B, Harbour D, Pegadiotes J, Natale J, Hamline M, Siefkes H. Protocol-Driven Initiation and Weaning of High-Flow Nasal Cannula for Patients With Bronchiolitis: A Quality Improvement Initiative. Pediatr Crit Care Med. 2023 Feb 1;24(2):112-122. doi: 10.1097/PCC.0000000000003136. Epub 2022 Dec 16. PMID 36661418
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Kepreotes E, Whitehead B, Attia J, Oldmeadow C, Collison A, Searles A, Goddard B, Hilton J, Lee M, Mattes J. High-flow warm humidified oxygen versus standard low-flow nasal cannula oxygen for moderate bronchiolitis (HFWHO RCT): an open, phase 4, randomised controlled trial. Lancet. 2017 Mar 4;389(10072):930-939. doi: 10.1016/S0140-6736(17)30061-2. Epub 2017 Feb 2. PMID 28161016
- [Background] Franklin D, Babl FE, Schlapbach LJ, Oakley E, Craig S, Neutze J, Furyk J, Fraser JF, Jones M, Whitty JA, Dalziel SR, Schibler A. A Randomized Trial of High-Flow Oxygen Therapy in Infants with Bronchiolitis. N Engl J Med. 2018 Mar 22;378(12):1121-1131. doi: 10.1056/NEJMoa1714855. PMID 29562151
- [Background] Collins C, Chan T, Roberts JS, Haaland WL, Wright DR. High-Flow Nasal Cannula in Bronchiolitis: Modeling the Economic Effects of a Ward-Based Protocol. Hosp Pediatr. 2017 Jul 25:hpeds.2016-0167. doi: 10.1542/hpeds.2016-0167. Online ahead of print. PMID 28743698
- [Background] Treasure JD, Hubbell B, Statile AM. Enough Is Enough: Quality Improvement to Deimplement High-Flow Nasal Cannula in Bronchiolitis. Hosp Pediatr. 2021 Apr;11(4):e54-e56. doi: 10.1542/hpeds.2021-005849. Epub 2021 Mar 22. No abstract available. PMID 33753361
- [Background] Franklin D, Schibler A. Rising Intensive Care Costs in Bronchiolitis Infants-Is Nasal High Flow the Culprit? Pediatr Crit Care Med. 2022 Mar 1;23(3):218-222. doi: 10.1097/PCC.0000000000002900. No abstract available. PMID 35238842
- [Background] Charvat C, Jain S, Orenstein EW, Miller L, Edmond M, Sanders R. Quality Initiative to Reduce High-Flow Nasal Cannula Duration and Length of Stay in Bronchiolitis. Hosp Pediatr. 2021 Apr;11(4):309-318. doi: 10.1542/hpeds.2020-005306. Epub 2021 Mar 22. PMID 33753362
- [Background] Peterson RJ, Hassumani DO, Hole AJ, Slaven JE, Tori AJ, Abu-Sultaneh S. Implementation of a High-Flow Nasal Cannula Management Protocol in the Pediatric ICU. Respir Care. 2021 Apr;66(4):591-599. doi: 10.4187/respcare.08284. Epub 2020 Sep 11. PMID 32917844